CLINICAL TRIAL: NCT04608838
Title: An Exploratory, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety and Efficacy of JTR-161 in Patients With Acute Ischemic Stroke
Brief Title: A Randomized Placebo-controlled Multicenter Trial to Evaluate the Efficacy and Safety of JTR-161, Allogeneic Human Dental Pulp Stem Cell, in Patients With Acute Ischemic stRoke (J-REPAIR)
Acronym: J-REPAIR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teijin Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JTR-161-201
Record Dates: First submitted 2020-09-08; First posted 2020-10-29 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Some care providers who involved in the preparation or administration of dosing solutions are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JTR-161 (Experimental)
  Interventions: Biological: JTR-161
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: JTR-161 — JTR-161 (1 or 3 × 10^8 cells/subject) will be suspended and administered in an intravenously infusion.
  Arms: JTR-161
Biological: Placebo — Placebo will be suspended and administered in an intravenously infusion.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a single intravenous administration of JTR-161 (allogeneic stem cell product derived from the dental pulp of healthy adult humans) to patients with acute ischemic stroke.

This study is comprised of 3 cohorts and conducted in the order of Cohort 1, Cohort 2 and Cohort 3.

Cohort 1 Arm-1: JTR-161, 1 × 10^8 cells/subject, 6 subjects Arm-2: Placebo, 2 subjects

The Data and Safety Monitoring Board (DSMB) and the Sponsor will decide whether Cohort 2 can be initiated or not.

Cohort 2 Arm-1: JTR-161, 3 × 10^8 cells/subject, 6 subjects Arm-2: Placebo, 2 subjects

DSMB and the Sponsor will decide whether Cohort 3 can be initiated or not and the dose of JTR-161 in Cohort 3.

Cohort 3 Arm-1: JTR-161, 1 × 10^8 cells/subject or 3 × 10^8 cells/subject, 30 subjects Arm-2: Placebo, 30 subjects

ELIGIBILITY:
Inclusion Criteria:

* Patients who have ischemic strokes in the anterior circulation
* Patients whose mRS is 0 or 1 prior to the onset of ischemic stroke
* Patients whose NIHSS score of ≥5 to ≤20 at screening
* Patients who can be administered dosing solutions within 48 h of stroke onset

Exclusion Criteria:

* Patients who have new ischemic lesion in the cerebellum or brainstem
* Patients whose consciousness level drops severely
* Patients whose infarct area is widespread
* Patients who have a clinically significant hemorrhagic transformation
* Patients who had seizures after onset of ischemic stroke
* Patients who have medical history of a neurological event such as stroke or clinically significant head trauma within 180 days prior to giving informed consent
* Patients who have poor blood pressure control
* Patients who have poor glycaemic control
* Patients who have one of the following complications

  1. Severe liver dysfunction
  2. Severe kidney dysfunction
  3. Severe heart failure
  4. Severe pulmonary dysfunction
* Patients who have severe infections
* Patients who have any neurological disorder affecting informed consent or study assessments
* Patients who have the malignant tumor, or medical history of malignant tumor within 2 years prior to the onset of ischemic stroke
* Patients who have a contraindication for MRI
* Patients who have thrombocytopenia
* Patients who have medical history of allergy to products derived from human tissues, bovine or porcine
* Patients who have medical history of allergy to streptomycin
* Patients who have undergone splenectomy in the past
* Patients who have a possibility of transient ischemic attack
* Patients who are scheduled to undergo revascularization (carotid endarterectomy, stent placement etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who achieved Excellent outcome (modified Rankin Scale [mRS] ≤1 and National Institutes of Health Stroke Scale [NIHSS] ≤1 and Barthel Index [BI] ≥95) on Day 91 in Cohort 3. | 91 days

SECONDARY OUTCOMES:
Percentage of patients who achieved mRS ≤ 1 or mRS ≤ 2 | 366 days
Percentage of patients who achieved BI ≥ 95 | 366 days
Percentage of patients who achieved NIHSS ≤ 1, who achieved improvement of ≥ 75%, and who achieved improvement of ≥ 10 points | 91 days
Changes in EQ-5D-5L scores | 366 days
  The EuroQOL 5 dimension 5-level (EQ-5D-5L) consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1="no problems", 2="slight problems", 3="moderate problems", 4="severe problems" and 5="extreme problems".
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Percentage of patients who achieved excellent outcome (mRS ≤ 1, NIHSS ≤ 1, and BI ≥ 95) | 91 days
Percentage of patients who showed overall improvement (mRS ≤ 2, NIHSS improvement of ≥ 75%, and BI ≥ 95) | 91 days
Incidence of Adverse events (signs and symptoms) | 366 days
Changes in Laboratory tests (hematology, blood chemistry, blood coagulation test, urinalysis) | 366 days
  Number of participants with clinical laboratory abnormalities for each parameter
  * hematology Red blood cell count, Hemoglobin, Hematocrit, Platelet count, Leukocyte count, Leukocyte formula (neutrophils, lymphocytes, monocytes, eosinophils, basophils)
  * blood chemistry Total protein, Albumin, Total bilirubin, Aspartate aminotransferase , Alanine aminotransferase, Alkaline phosphatase , Lactate dehydrogenase , γ-Glutamyltransferase, Blood urea nitrogen , Creatinine, Uric acid, Sodium, Potassium, Calcium, Chloride, Creatine kinase , C-reactive protein
  * blood coagulation Prothrombin time (International normalized ratio) , Activated partial thromboplastin time
  * urinalysis Urine Protein, Urine Glucose
Changes in Vital signs (blood pressure [systolic/diastolic], pulse rate, body temperature) | 366 days
  Number of participants of the vital signs abnormalities for each parameter: blood pressure (mmHg), pulse rate (bpm) and body temperature (℃).
Changes in Oxygen saturation (SpO2) | 366 days
Changes in findings of imaging examination by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT). | 31 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Medical School Hospital, Bunkyo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suda S, Nito C, Ihara M, Iguchi Y, Urabe T, Matsumaru Y, Sakai N, Kimura K; J- REPAIR trial group. Randomised placebo-controlled multicentre trial to evaluate the efficacy and safety of JTR-161, allogeneic human dental pulp stem cells, in patients with Acute Ischaemic stRoke (J-REPAIR). BMJ Open. 2022 May 24;12(5):e054269. doi: 10.1136/bmjopen-2021-054269. PMID 35613802